CLINICAL TRIAL: NCT00057096
Title: Onsite Versus Referral Models of Primary Care for Substance Abusing Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUI 99-109
Record Dates: First submitted 2003-03-27; First posted 2003-03-28 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Substance Abuse; Primary Medical Care
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: On-site vs. referral methods of care

INTERVENTIONS:
Procedure: On-site vs. referral methods of care

SUMMARY:
Veterans presenting for treatment of substance use disorders (SUDs) often have multiple and serious comorbid medical conditions that affect functional health status and health care costs. Prior studies show higher rates of medical follow-up when onsite primary health care was provided to patients with SUDs within an addictions clinic (onsite care). However, no data are available on differences between onsite versus referral models of primary care delivery in terms of clinical outcomes and total health care costs.

DETAILED DESCRIPTION:
Background:

Veterans presenting for treatment of substance use disorders (SUDs) often have multiple and serious comorbid medical conditions that affect functional health status and health care costs. Prior studies show higher rates of medical follow-up when onsite primary health care was provided to patients with SUDs within an addictions clinic (onsite care). However, no data are available on differences between onsite versus referral models of primary care delivery in terms of clinical outcomes and total health care costs.

Objectives:

The objectives of this study are to compare patients with SUDs who receive onsite primary care in a VA outpatient addictions clinic to those referred for primary care to the general internal medicine clinic on: 1) medical outcomes and quality of life; 2) SUD treatment outcomes; and 3) overall health care costs. This information will assist in identifying practice guidelines for providing preventive services and treatment for acute and chronic medical conditions to individuals in SUD treatment.

Methods:

This study is a randomized clinical trial with two treatment conditions: 1) onsite primary care in the Addictions Treatment Center (ATC; experimental); or 2) referral primary care in the General Internal Medicine Clinic (GIMC; control). Subjects are assessed at baseline and at 3, 6, and 12-month time points. The sample includes 720 veterans, newly presenting or returning to SUD treatment, who exhibited a chronic medical condition at screening, did not have a primary care provider; and did not present with a serious medical condition requiring ongoing care in three or more organ systems. Medical status outcome measures include scores on the SF-36, and total emergency room visits and medical or surgical inpatient admissions. Substance abuse outcomes are measured by treatment retention, changes in Addiction Severity Index (ASI) scores, and self-reported alcohol use. Lastly, overall VA health care costs per subject per the 12-month period following randomization are compared across groups. The main analysis involves intent-to-treat analysis of group (onsite vs. referral) by time (3, 6, 12-month) using random effects regression models.

Status:

Complete. All subjects completed study interventions as of 3/31/2004. Currently data analysis is ongoing.

ELIGIBILITY:
Inclusion Criteria:

Enrolling in addictions treatment, has no primary care provider currently and has some ongoing medical concern that would benefit from primary care.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Saxon, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

REFERENCES:
- [Result] Saxon AJ, Malte CA, Sloan KL, Baer JS, Calsyn DA, Nichol P, Chapko MK, Kivlahan DR. Randomized trial of onsite versus referral primary medical care for veterans in addictions treatment. Med Care. 2006 Apr;44(4):334-42. doi: 10.1097/01.mlr.0000204052.95507.5c. PMID 16565634
- [Result] Davis TM, Carpenter KM, Malte CA, Carney M, Chambers S, Saxon AJ. Women in addictions treatment: comparing VA and community samples. J Subst Abuse Treat. 2002 Jul;23(1):41-8. doi: 10.1016/s0740-5472(02)00242-8. PMID 12127467
- [Result] Saxon A, Sloan K, Nichol P, Howell D, Bush K, Calsyn D, Baer J, Felker B, Kivlahan D. Substance Dependent Individuals Often Lack Awareness of Their Medical Conditions. Drug and Alcohol Dependence. 2002 Oct 15; 66:S156-S156.
- [Result] Calsyn DA, Saxon AJ, Bush KR, Howell DN, Baer JS, Sloan KL, Malte CA, Kivlahan DR. The Addiction Severity Index medical and psychiatric composite scores measure similar domains as the SF-36 in substance-dependent veterans: concurrent and discriminant validity. Drug Alcohol Depend. 2004 Nov 11;76(2):165-71. doi: 10.1016/j.drugalcdep.2004.04.018. PMID 15488340
- [Result] Zarkin GA, Bray JW, Mitra D, Cisler RA, Kivlahan DR. Cost methodology of COMBINE. J Stud Alcohol Suppl. 2005 Jul;(15):50-5; discussion 33. doi: 10.15288/jsas.2005.s15.50. PMID 16223056
- [Result] Saxon A, Calsyn D, Sloan K, Baer J, Kivlahan D, Felker B, Nichol P, Paden G, DeMarco F. Primary care attendance of substance dependent patients. Drug and Alcohol Dependence. 2001 Jun 1; 63:S1.
- [Result] Caldeiro RM, Malte CA, Calsyn DA, Baer JS, Nichol P, Kivlahan DR, Saxon AJ. The association of persistent pain with out-patient addiction treatment outcomes and service utilization. Addiction. 2008 Dec;103(12):1996-2005. doi: 10.1111/j.1360-0443.2008.02358.x. Epub 2008 Oct 8. PMID 18855809
- [Result] Buchholz JR, Malte CA, Calsyn DA, Baer JS, Nichol P, Kivlahan DR, Caldeiro RM, Saxon AJ. Associations of housing status with substance abuse treatment and service use outcomes among veterans. Psychiatr Serv. 2010 Jul;61(7):698-706. doi: 10.1176/ps.2010.61.7.698. PMID 20592005